CLINICAL TRIAL: NCT04055155
Title: Discovering the Capacity of Primary Care Frontline Staff to Deliver a Low-Intensity Technology-Enhanced Intervention to Treat Geriatric Depression
Brief Title: Technology-enabled Task-sharing for Depression in Primary Care
Status: Withdrawn | Type: Observational
Why Stopped: Pandemic halt
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Oleg Zaslavsky, Assistant Professor, Biobehavioral Nursing and Health Systems, University of Washington
Other Study IDs: STUDY00006748; P50MH115837 (NIH)
Record Dates: First submitted 2019-08-09; First posted 2019-08-13 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Depression; Depression in Old Age
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Staff/Provider end-users: Testing usability of a technology-enabled behavioral intervention for depression among provider end-users in primary care.
- Patient participants: Testing acceptability, feasibility, and preliminary effectiveness of a technology-enabled behavioral intervention for depression among patients with depression in primary care.

SUMMARY:
This study will explore and test the feasibility, acceptability, usability, and preliminary effectiveness of a technology-enabled intervention for depression using task-sharing in primary care. We will a) discover barriers and facilitators to task-sharing by frontline primary care staff; b) design an implementation strategy to support task-sharing to deliver a technology-enabled intervention for depression; and c) conduct a small open-label usability trial of the technology-enabled intervention for depression.

DETAILED DESCRIPTION:
Older adults with depression typically present to primary care rather than specialty mental health treatment and are often un- or undertreated, as the demand for mental health services is greater than the supply of trained providers. Technology is one method to improve access to care by making evidence-based psychosocial interventions (EBPIs) readily accessible. A second method comes from global mental health research, demonstrating that task-sharing can equip non-specialists to provide effective mental health care. This study combines these two approaches, exploring how technology-enhanced EBPI could be used by frontline primary care staff (e.g., nurses, medical assistants) to expand workforce capacity to deliver acceptable, sustainable, and effective treatment for depression. Specifically, we will use task-sharing to deliver a mobile Motivational Physical Activity Targeted Intervention (MPATI), which is based on behavioral activation for depression and uses wearable accelerometer technology to trigger personalized activity goal monitoring. This proposal uses the Discover, Design/Build, Test (DDBT) framework, which leverages user-centered design and implementation science to discover implementation barriers to using task-sharing to deliver MPATI in primary care, to design an implementation strategy to support MPATI delivery, and to conduct a pilot usability trial to test the implementation strategy with the most suitable frontline staff.

ELIGIBILITY:
Inclusion Criteria:

Clinics:

1. have at least 1 full-time registered nurse (RN) and/or medical assistant (MA) on staff
2. include older adults on their patient panels.

Clinic administrators

1. have an administrative or leadership role in the clinic
2. have been employed in their current role for at least 6 months.

Frontline staff

1. provide care as RN, MA, case manager, behavioral health consultant, or similar role identified by Practice Champion
2. be employed at the participating clinic for at least 6 months.

Patients

1. be ≥65 years of age
2. report moderate to moderately severe depressive symptoms based on a PHQ-9 score of 10-20
3. own or have access to a smartphone
4. have internet or cellular data plan
5. receive medical clearance from their primary care provider to participate in unstructured physical activity.

Patient exclusion criteria will be based on medical chart review by Practice Champion and include:

1. current suicidality
2. severe vision or hearing impairment
3. pronounced cognitive impairment
4. use of assistive devices that would impede physical activity.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinics: administrators, primary care providers, behavioral health providers, frontline primary care staff (e.g., nurses, medical assistants)
  Patients: older adult primary care patients with mild-to-moderate depressive symptoms
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Usability (system usability scale) | after 2 week usability trial
  usability of MPATI intervention among provider end-users
Usability (qualitative interviews) | after 2 week usability trial
  usability of MPATI intervention among provider end-users

SECONDARY OUTCOMES:
feasibility -- patient recruitment | end of pilot trial (2 weeks per patient)
  feasibility of MPATI intervention for geriatric depression in primary care
acceptability -- patient retention | end of pilot trial (2 weeks per patient)
  acceptability of MPATI intervention for geriatric depression in primary care
depressive symptoms (patient) | pre-post 2 week pilot trial
  Patient Health Questionnaire (PHQ-9) total scores to assess depressive symptoms (total score range 0-27; higher scores reflect greater depressive symptoms)
functioning (patient) | pre-post 2 week pilot trial
  Sheehan Disability Scale (SDS) total scores to assess functional impairment; total scores range from 0 (unimpaired) to 30 (highly impaired).

OTHER OUTCOMES:
user burden | end of 2 week pilot trial
  user burden of technology-enabled intervention for patients and providers

CONTACTS AND LOCATIONS:
Overall Officials: Oleg Zaslavsky, PhD, Principal Investigator — University of Washington; Brenna Renn, PhD, Principal Investigator — University of Washington
Locations (1):
- Univeristy of Washington, Seattle, Washington, United States